CLINICAL TRIAL: NCT01369199
Title: Combination Entecavir and Peginterferon Therapy in HBeAg-Positive Immune-Tolerant Adults With Chronic Hepatitis B
Acronym: HBRN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of Pittsburgh (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK082864 HBRN IT Adult Trial; U01DK082916 (NIH); U01DK082843 (NIH); U01DK082863 (NIH); U01DK082864 (NIH); U01DK082866 (NIH); U01DK082867 (NIH); U01DK082871 (NIH); U01DK082872 (NIH); U01DK082874 (NIH); U01DK082919 (NIH); U01DK082923 (NIH); U01DK082927 (NIH); U01DK082943 (NIH); U01DK082944 (NIH); P30DK050306 (NIH); A-DK-3002-001 (Other Grant/Funding Number: Interagency agreement with NIDDK); M01RR000040 (NIH); UL1TR000058 (NIH); UL1TR000004 (NIH); UL1TR001111 (NIH); UL1RR024986 (NIH); NCT01534611 (obsolete NCT alias)
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Immune-tolerant hepatitis B; HBV
MeSH Terms: conditions — Hepatitis B | interventions — entecavir; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Peginterferon and entecavir (Experimental): A combination of 8 weeks of entecavir followed by 40 weeks of both entecavir and peginterferon.
  Interventions: Drug: Entecavir and peginterferon

INTERVENTIONS:
Drug: Entecavir and peginterferon — Entecavir 0.5 mg daily orally for 48 weeks plus peginterferon 180 µg sq weekly during weeks 9-48 of treatment.
  Other Names: PEGASYS, peginterferon alfa 2a, Baraclude

SUMMARY:
The investigators evaluated the safety and efficacy of a short lead-in course (8 weeks) of entecavir followed by combination of entecavir plus peginterferon alfa-2a for 40 weeks.

DETAILED DESCRIPTION:
To determine the efficacy of treatment with 8 weeks of entecavir followed by 40 weeks of both entecavir and peginterferon in the treatment of chronic hepatitis B in hepatitis B "e" antigen (HBeAg) positive adults who are in the immune tolerant phase.

To evaluate safety and sustained responses after treatment with entecavir and peginterferon alfa-2a in the treatment of chronic hepatitis B in HBeAg positive adults who are in the immune tolerant phase.

A single arm treatment study of 8 weeks of entecavir followed by 40 weeks of both entecavir and peginterferon alfa-2a in adults with HBeAg-positive chronic hepatitis B with normal or near normal alanine aminotransferase (ALT) levels and high serum levels of hepatitis B virus (HBV) DNA ("immune tolerant" HBeAg-positive chronic hepatitis B). All participants followed for 48 weeks after treatment discontinuation (week 96 for those who completed treatment).

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in & completed the baseline evaluation for NCT01263587 or completed the necessary components of NCT01263587 by the end of baseline visit.
* >18 years of age at the baseline visit (day 0). Patients >50 years of age at baseline will need to have a liver biopsy as standard of care with hepatic activity index (HAI) ≤3 & Ishak fibrosis score ≤1 within 96 weeks prior to baseline visit.
* Documented chronic HBV infection as evidenced by detection of HBsAg in serum for ≥24 weeks prior to baseline visit OR at least one positive HBsAg & negative anti-hepatitis B core (HBc) immunoglobulin (IgM) within 24 weeks prior to baseline visit OR at least one positive HBsAg & two positive HBV DNA over a period of ≥24 weeks prior to baseline visit.
* Presence of HBeAg in serum at last screening visit within 6 weeks of baseline visit.
* Serum HBV DNA level >10˄7 IU/mL on at least two occasions at least 12 weeks apart during the 52 weeks before baseline visit. One of the two HBV DNA levels must be within 6 weeks of baseline visit.
* ALT levels persistently ≤45 U/L in males, ≤30 U/L in females (approx. 1.5 times the upper limit of normal (ULN) range) as documented by at least three values: one taken 28-52 weeks before baseline visit, one taken 6 to 24 weeks before the baseline visit, & the final value within 6 weeks prior to baseline visit.
* No evidence of hepatocellular carcinoma (HCC) based upon alpha-fetoprotein (AFP) ≤20 ng/mL at screening visit (up to 6 weeks prior to baseline visit). a. Participants who meet American Association for the Study of Liver Diseases (AASLD) criteria for HCC surveillance must have negative liver imaging as shown by ultrasound, computerized tomography (CT) or magnetic resonance imaging (MRI) within 28 weeks prior to baseline visit. b. Participants with AFP >20 ng/mL must be evaluated clinically with additional imaging & shown not to have HCC on CT or MRI before they can be enrolled.

Exclusion Criteria:

* History of hepatic decompensation
* Evidence of decompensated liver disease prior to or during screening, including direct bilirubin >0.5 mg/dL, international normalization ratio (INR) >1.5, or serum albumin <3.5 g/dL.
* Platelet count <120,000/mm3, hemoglobin <13 g/dL (males) or <12 g/dL (females), absolute neutrophil count < 1500 /mm3 (<1000/mm3 for African-Americans) at last screening visit.
* Previous treatment with medications that have established activity against HBV including interferon & nucleos(t)ide analogs ≥24 weeks. Patients with <24 weeks of prior HBV treatment & a wash-out period >24 weeks are not excluded.
* Known allergy or intolerance to study medications.
* Females who are pregnant or breastfeeding. Females of childbearing potential unable or unwilling to use a reliable method of contraception during the treatment period.
* Renal insufficiency with calculated creatinine clearance <50 mL/min at screening.
* History of alcohol or drug abuse within 48 weeks of baseline visit.
* Previous liver or other organ transplantation (including engrafted bone marrow).
* Any other concomitant liver disease, including hepatitis C or D. Non-alcoholic fatty liver disease (NAFLD) with steatosis &/or mild to moderate steatohepatitis is acceptable but NAFLD with severe steatohepatitis is exclusionary.
* Presence of anti-hepatitis D virus (HDV) or anti-hepatitis C virus (HCV) (unless HCV RNA negative) in serum on any occasion in the 144 weeks prior to baseline visit. Presence of anti-HIV (test completed within 6 weeks prior to baseline visit).
* Pre-existing psychiatric condition(s), including, but not limited to: current moderate or severe depression, history of depression requiring hospitalization within the past 10 years, history of suicidal or homicidal attempt within the past 10 years, history of severe psychiatric disorders as determined by a study physician.
* History of immune-mediated or cerebrovascular disease, chronic pulmonary or cardiac disease associated with functional limitation, retinopathy, uncontrolled thyroid disease, poorly controlled diabetes or uncontrolled seizure disorder, as determined by a study physician.
* Any medical condition that would, in the opinion of a study physician, be predicted to be exacerbated by therapy or that would limit study participation.
* Any medical condition requiring, or likely to require, chronic systemic administration of corticosteroids or other immunosuppressive medications during the course of this study.
* Evidence of active or suspected malignancy, or a history of malignancy within the 144 weeks prior to baseline visit (except adequately treated carcinoma in situ or basal cell carcinoma of the skin).
* Expected need for ongoing use of any antivirals with activity against HBV during the course of the study.
* Concomitant use of complementary or alternative medications purported to have antiviral activity.
* Participation in any other clinical trial involving investigational drugs within 30 days of the baseline visit or intention to participate in another clinical trial involving investigational drugs during participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-05; Primary Completion 2017-02-14 (Actual); Study Completion 2017-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Averell Sherker, MD, Study Chair — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Anna Lok, MD, Principal Investigator — University of Michigan
Locations (21):
- United States (20):
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Queen's Medical Center, Honolulu, Hawaii
  - NIH Clinical Center, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All data collected will be sent to the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)-supported data repository.
Supporting Information: Study Protocol, SAP
Time Frame: At completion of HBRN project. Length of availability determined by NIDDK data repository.
Access Criteria: Per NIDDK-supported data repository

REFERENCES:
- See also: Click here for more information about the Hepatitis B Research Network — http://www.hepbnet.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-eight (28) adults were enrolled at 11 clinical sites in the United States and Canada between 12/18/12 and 04/29/15.
Groups:
- Peginterferon and Entecavir: Entecavir 0.5 mg daily orally for 48 weeks plus peginterferon alfa-2a 180 μg subcutaneously weekly during weeks 9-48 of treatment. After treatment discontinuation, follow-up for 48 weeks.
Period: Overall Study
Arm/Group | Peginterferon and Entecavir
Started | 28
End of Treatment (EOT) | 26 (1 withdrew consent before treatment,1 missed end of treatment (EOT) visit but completed follow-up.)
Completed (End of follow-up) | 25
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- Peginterferon and Entecavir: Entecavir 0.5 mg daily orally for 48 weeks plus peginterferon alfa-2a 180 μg subcutaneously weekly during weeks 9-48 of treatment. After treatment discontinuation, follow-up off treatment for 48 weeks.
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 37.2 [22.2 to 61.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 27
  Black/African American | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 9
  United States | 19
Hepatitis B Virus (HBV) DNA [Median (Full Range); unit: log10 IU/mL] | 8.2 [7.2 to 8.8]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With HBeAg Loss (Lack of Detectable HBeAg) AND HBV DNA ≤1,000 IU/mL
Description: Lack of data was considered to be treatment failure.
Time Frame: End of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | 0 [0 to .123]

2. Primary Outcome: Incidence of Adverse Events (AEs) Per Person-Year of Observation
Description: The number of AEs includes both AEs and Serious Adverse Events (SAEs). The incidence is calculated as the number of AEs divided by the number of person-years of observation, which is the sum, across all participants, of the number of years between the start of treatment and the end of treatment, or the end of follow-up, respectively.
Time Frame: From first treatment to the end of treatment (up to 48 weeks) and the end of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Events per person-year of observation
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Events per person-year of observation
  End of treatment (Up to 48 weeks) | 1.60 [1.17 to 2.19]
  End of follow-up (Up to 96) weeks | 0.86 [0.64 to 1.17]

3. Primary Outcome: Incidence of Serious Adverse Events (SAEs) Per Person-Year
Description: The incidence is calculated as the number of SAEs divided by the number of person-years of observation, which is the sum, across all participants, of the number of years between the start of treatment and the end of treatment, or the end of follow-up, respectively.
Time Frame: From first treatment to the end of treatment (up to 48 weeks) and the end of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: SAEs per person-year of observation
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
SAEs per person-year of observation
  End of treatment (Up to 48 weeks) | 0 [NA to NA] — 95% Confidence Interval (CI) around 0 not calculated
  End of follow-up (Up to 96 weeks) | .021 [.003 to .146]

4. Secondary Outcome: Proportion of Participants With HBeAg Loss
Time Frame: End of treatment (up to 48 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | .036 [.001 to .183]

5. Secondary Outcome: Proportion of Participants With HBeAg Loss
Time Frame: End of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | .036 [.001 to .183]

6. Secondary Outcome: Proportion of Participants With HBeAg Seroconversion
Time Frame: End of treatment (up to 48 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | .036 [.001 to .183]

7. Secondary Outcome: Proportion of Participants With HBeAg Seroconversion
Time Frame: End of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | .036 [.001 to .183]

8. Secondary Outcome: Proportion of Participants With HBsAg Loss
Time Frame: End of treatment (up to 48 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | 0 [0 to .123]

9. Secondary Outcome: Proportion of Participants With HBsAg Loss
Time Frame: End of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | 0 [0 to .123]

10. Secondary Outcome: Proportion of Participants With HBsAg Seroconversion
Time Frame: End of treatment (up to 48 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | 0 [0 to .123]

11. Secondary Outcome: Proportion of Participants With HBsAg Seroconversion
Time Frame: End of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | 0 [0 to .123]

12. Secondary Outcome: Proportion of Participants With Alanine Aminotransferase (ALT) <45 U/L for Men, <30 U/L for Women
Time Frame: End of treatment (up to 48 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | .571 [.245 to .628]

13. Secondary Outcome: Proportion of Participants With ALT <45 U/L for Men, <30 U/L for Women
Time Frame: End of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | .750 [.551 to .893]

14. Secondary Outcome: Proportion of Participants With ALT Normalization (Men <30 U/L, Women <20 U/L)
Time Frame: End of treatment (up to 48 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | .393 [.215 to .594]

15. Secondary Outcome: Proportion of Participants With ALT Normalization (Men <30 U/L, Women <20 U/L)
Time Frame: End of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | .464 [.275 to .661]

16. Secondary Outcome: Proportion of Participants With HBV DNA ≤1000 IU/mL
Time Frame: End of treatment (up to 48 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | .929 [.765 to .991]

17. Secondary Outcome: Proportion of Participants With HBV DNA ≤1000 IU/mL
Time Frame: End of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | 0 [0 to .123]

18. Secondary Outcome: Proportion of Participants With HBV DNA <20 IU/mL
Time Frame: End of treatment (up to 48 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | .179 [.061 to .369]

19. Secondary Outcome: Proportion of Participants With HBV DNA <20 IU/mL
Time Frame: End of follow-up (up to 96 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | 0 [0 to .123]

20. Secondary Outcome: Absence of Detectable Antiviral Drug-resistance HBV Mutations
Description: HBV drug resistance variant testing was performed at the CDC laboratory. The sequences of the HBV polymerase spanning nucleotide positions 311-1021 were determined by Sanger sequencing. Drug resistance mutations that were tested in this study included L80VI, L82M, T128N, W153Q, F166L, I169T, V173L, L180M, A181TV, T184ACFGILMS, V191T, A194T, A200V, S202ETV, M204IV, V207I, N236T, M250ILV, and G145R.
Time Frame: End of treatment (up to 48 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Peginterferon and Entecavir
Number analyzed (Participants) | 28
Proportion of participants | .893 [.718 to .977]

ADVERSE EVENTS:
Time Frame: Study entry (consent) to the end of follow-up (up to 96 weeks after treatment initiation).
Description: Asked at each visit. Expected symptoms/signs or common side effects of meds not reported (these are termed Adverse Effects). Below is a guide for recording adverse events which are at the discretion of the investigator.
  1. Symptom or event requiring discontinuation of study medication.
  2. New symptom or event requiring a written prescription for treatment.
  3. New symptom or event resulting in a referral to another provider.
  4. Grade 3 or 4 event per the NCI Common Toxicity Criteria.
Groups:
- Peginterferon and Entecavir: Entecavir 0.5 mg daily orally for 48 weeks plus peginterferon alfa-2a 180 μg subcutaneously (sq) weekly during weeks 9-48 of treatment. After treatment discontinuation, follow-up off treatment will be for 48 weeks.
Arm/Group | Peginterferon and Entecavir
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 1/28
Other Adverse Events (participants affected / at risk) | 14/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon and Entecavir (N=28)
Malaria (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon and Entecavir (N=28)
Low white blood cells, platelets, and absolute neutrophil count (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Altered thyroid function (Endocrine disorders) | 1 (1)
Graves disease (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1)
Heartburn and diarrhea (Gastrointestinal disorders) | 1 (1)
Poor appetite (Gastrointestinal disorders) | 1 (1)
Upset stomach (Gastrointestinal disorders) | 1 (1)
Decrease in appetite (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Head cold (General disorders) | 1 (1)
Sore throat (General disorders) | 1 (1)
Swollen lips (General disorders) | 1 (1)
Upper respiratory infection (General disorders) | 1 (1)
Infection in right forefinger (Infections and infestations) | 1 (1)
Intermittent finger joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Shingles (Nervous system disorders) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1)
Depressive disorder (Psychiatric disorders) | 1 (1)
Foul urine smell (Renal and urinary disorders) | 1 (1)
Frequent urination - prophylaxis (Renal and urinary disorders) | 1 (1)
Penile yeast infection (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 2 (4)
Pneumococcal pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Hair loss) (Skin and subcutaneous tissue disorders) | 3 (4)
Bruising on legs (Skin and subcutaneous tissue disorders) | 1 (1)
Hives (Skin and subcutaneous tissue disorders) | 1 (1)
Itchiness at injection site (intermittent) (Skin and subcutaneous tissue disorders) | 1 (1)
Rash and itchiness on lower jaw (Skin and subcutaneous tissue disorders) | 1 (1)
Redness at injection site (Skin and subcutaneous tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Early termination of recruitment per Data and Safety Monitoring Board.

1 case with multiple central and local lab discrepancies was not considered to have HBeAg loss since central lab was always negative.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
From the Publications and Presentations policy "Disagreements between the HBRN Steering Committee and the NIDDK on the merits of journal submission of a specific manuscript will be mediated through discussion on Steering Committee conference calls, ad hoc conference calls or during face to face Steering Committee meetings. The decision of the NIDDK is final and cannot be appealed."

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-08-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT01369199/Prot_SAP_000.pdf